CLINICAL TRIAL: NCT04957017
Title: Effect of Training on Given to Women With Chronic Disease on Hand-Washing Behaviours, Attitudes and Nutrition During the Covid-19 Pandemic
Brief Title: Effect of Hand-Washing Training in Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Nurten Terkes, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GO 2020/192
Record Dates: First submitted 2021-07-04; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Chronic Disease; Covid-19 Pandemic
Keywords: COVID-19; hand hygiene; chronic disease
MeSH Terms: conditions — Chronic Disease; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The women with chronic disease were met, and the Descriptive Information Form, Social Hand-Washing Knowledge Form and the "Nutritional Knowledge Level Scale for Adults" were filled with the volunteer ones face-to-face at their homes, complying with the social distance rules before the training. After the data was collected, the women in the intervention group were trained on "Hand-Washing and Nutrition during the COVID-19 period". The training on hand-washing and nutrition was given using the "Hand-Washing and Nutrition Training Guide" prepared by the researchers, and the "Hand-Washing and Nutrition Training Manual" covering the content of the training, was distributed to the women at the end of the training. The data collection forms were re-filled three months after the training.
  Interventions: Behavioral: Training
- Control group (No Intervention): The women with chronic disease were met, and the Descriptive Information Form, Social Hand-Washing Knowledge Form and the Nutritional Knowledge Level Scale for Adults were filled face-to-face at their homes with the ones volunteering to participate in the study, complying with the social distance rules. The same survey was re-filled after three months. No training was given to the women with chronic disease during the three-month period. After the research was completed, a 45 minute-training which is the same with the one provided to the intervention group was given individually to the control group, complying the social distance rules.

INTERVENTIONS:
Behavioral: Training — After the data was collected, the women in the intervention group were trained on "Hand-Washing and Nutrition during the COVID-19 period". The training on hand-washing and nutrition was given using the "Hand-Washing and Nutrition Training Guide" prepared by the researchers, and the "Hand-Washing and Nutrition Training Manual" covering the content of the training, was distributed to the women at the end of the training
  Arms: Intervention group

SUMMARY:
This study was conducted in order to inform, the women with chronic disease in rural areas, about hand-washing and nutrition, and to evaluate the efficiency of the training program. A randomized-controlled trial was performed based on CONSORT checklist. 90 women in total were included in the study, 45 for each group. The women in the intervention group were given, by the researcher, the training on the importance of hand-washing and appropriate food choices. The training given to the women in rural areas created significant benefit for them to have the appropriate food choices and hand-washing behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Be women, agreeing to participate.

Exclusion Criteria:

* Be man, unable to communicate.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
The Nutritional Knowledge Level Scale for Adults (NKLSA) | Three months
  The Nutritional Knowledge Level Scale for Adults (NKLSA) developed by Batmaz in 2018 and whose validity and reliability were studied, the 20 statements under the heading "Basic Nutritional and Food-Health Knowledge" and 12 statements under the heading "Food Choice" were responded using one of the following: strongly agree, agree, neither agree nor disagree, disagree, and strongly disagree. The participants who responded the inappropriate statements by "strongly agree" got 0 point; those who "agreed" with these statements got 1 point; those who neither agreed nor disagreed got 2 points; those who disagreed got 3 points, and those who strongly disagreed with them got 4 points. The maximum score that can be obtained from the "Basic Nutritional and Food-Health Knowledge" is 80, and the maximum score to be obtained from the "Food Choice" is 48.
Social Hand-Washing Knowledge Form | Three months
  Social Hand-Washing Knowledge Form was created by the researchers by scanning the literature (Kilpatrick et al., 2018; Lynch et al., 2020; Wu et al., 2013), and the authors received expert opinions from 3 academic members for the content validity of the knowledge statements. The answers given to the questions were scored as No "0", Occasionally "1", Yes "2". Question 11 included in the investigators survey was reversely scored. The lowest score to be obtained from the investigators survey was 0 and the highest score was 22. As the investigators considered it more comprehensible to convert this score into a hundred scale and make the investigators evaluations over 100 points, the investigators evaluated the total score obtained by each case through converting it into a hundred scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy university, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
There is not plan.

REFERENCES:
- [Background] Geleta TA, Deriba BS, Beyane RS, Mohammed A, Birhanu T, Jemal K. COVID-19 Pandemic Preparedness and Response of Chronic Disease Patients in Public Health Facilities. Int J Gen Med. 2020 Nov 5;13:1011-1023. doi: 10.2147/IJGM.S279705. eCollection 2020. PMID 33177864
- [Result] Cintoni M, Rinninella E, Annetta MG, Mele MC. Nutritional management in hospital setting during SARS-CoV-2 pandemic: a real-life experience. Eur J Clin Nutr. 2020 May;74(5):846-847. doi: 10.1038/s41430-020-0625-4. Epub 2020 Apr 6. No abstract available. PMID 32253375